CLINICAL TRIAL: NCT00977821
Title: Embryo Developmental Capacity After Egg Banking in an Ovum Donation Program
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Principal Investigator, Carlos Simon, Dr. Carlos Simon MD PhD, Instituto Valenciano de Infertilidad, IVI VALENCIA
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 0901-F-054-CS
Record Dates: First submitted 2009-09-15; First posted 2009-09-16 (Estimated); Last update posted 2015-04-22 (Estimated); Status verified 2015-04

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- fresh (Active Comparator): Embryo transfer with fresh oocytes
  Interventions: Other: IVF
- Frozen (Experimental): Embryo transfer with vitrified oocytes
  Interventions: Other: Oocyte Vitrification

INTERVENTIONS:
Other: IVF
  Arms: fresh
Other: Oocyte Vitrification
  Arms: Frozen

SUMMARY:
For an efficient "egg banking" system, an equally efficient cryopreservation strategy that ensures the viability of the oocytes is required. Very recently, improved and new methods are yielding satisfactory results. In particular, vitrification is providing excellent results for both survival and clinical outcomes. However, to evaluate the over all out come there are other parameters to be considered. In this sense, capacity development of embryos generated after oocyte vitrification is a major factor when assessing the viability of vitrified oocytes. Accordingly, the evaluation of the capacity of vitrified oocytes to reach the blastocyst stage will be highly valuable to fully assess the effectiveness of the "egg banking" and its contribution to ovum donation programs.

The aim of this study is to evaluate the developmental capacity of vitrified oocytes by their ability to reach the blastocyst stage. The study includes oocyte donation cycles conducted with vitrified versus fresh oocytes.

ELIGIBILITY:
Inclusion Criteria:

* 18-35 year old
* Normal response (8-15 follicles) to long protocol of ovarian stimulation with hCG
* Donors with normal menstrual cycles (21-35 day duration)
* Donors with BMI between 18-25 Kg/m2

Exclusion Criteria:

* Donors with two or more previous miscarriages
* Polycystic ovary syndrome
* Donors with antecedents of poor embrionary quality not attributed to masculine factor
* Donors with drop of estradiol of more than 10% or estradiol plateau.
* Donors with a high response>20 oocytes and or levels above 3000pg/ml of estradiol the day of the administration of chorionic gonadotrophin (hCG)

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 625 (Actual)
Dates: Start 2009-09; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Mean outcome measures will be survival, fertilization and blastocyst rates and clinical outcome. | 10 months

CONTACTS AND LOCATIONS:
Locations (1):
- IVI Valencia, Valencia, Spain